CLINICAL TRIAL: NCT03026907
Title: Efficacy of Oral Alitretinoin Versus Oral Azathioprine in Patients With Severe Chronic Non-hyperkeratotic Hand Eczema. A Randomized Prospective Open-label Trial With Blinded Outcome Assessment
Brief Title: Alitretinoin vs Azathioprine in Severe Non-hyperkeratotic Hand Eczema
Acronym: ALIAZ
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Marie-Louise A Schuttelaar, MD, PhD, Principal investigator, dermatologist, MD, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52232
Record Dates: First submitted 2016-08-18; First posted 2017-01-20 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Hand Eczema
Keywords: Alitretinoin; Azathioprine; Hand eczema
MeSH Terms: interventions — Alitretinoin; Azathioprine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alitretinoin (Active Comparator): Patients with severe chronic non-hyperkeratotic hand eczema, randomized to treatment with alitretinoin.
  Interventions: Drug: Alitretinoin
- Azathioprine (Active Comparator): Patients with severe chronic non-hyperkeratotic hand eczema, randomized to treatment with azathioprine.
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Alitretinoin — Oral alitretinoin capsule of 30mg once daily for a total of 24 weeks.
  Other Names: Toctino; 9-cis-retinoic acid; ATC code: D11AH04
  Arms: Alitretinoin
Drug: Azathioprine — Oral azathioprine tablets twice daily in a dose of 1.5 or 2.5mg/kg/day, depending on the thiopurine methyltransferase (TPMT) activity.
  Other Names: Imuran; Azafalk; ATC code: L04AX01
  Arms: Azathioprine

SUMMARY:
The purpose of this study is to compare the efficacy of alitretinoin and azathioprine in the treatment of patients with severe chronic non-hyperkeratotic hand eczema.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 75 years
* Severe or very severe chronic non-hyperkeratotic hand eczema for a minimum duration of 3 months as defined by a Physician Global Assessment (PGA) using a validated Photoguide
* Refractory to standard therapy, defined as:

Patients received treatment with topical corticosteroids of class II or higher for at least 8 weeks within 3 months before enrolment, with either no response or a transient response. Patients had also received standard skin care, including emollients and barrier protection as appropriate, without significant improvement. Patients had avoided irritants and allergens, if identified, without significant improvement.

* Women of childbearing potential are required to use at least two forms of contraception for at least 1 month before starting treatment, during treatment, and for at least 1 month after finishing treatment; these women are required to take monthly pregnancy tests
* Able to provide written Informed Consent
* Able to speak and read the Dutch language

Exclusion Criteria:

General criteria prior to randomization

* Treatment with alitretinoin or azathioprine in the previous 3 months
* Hyperkeratotic palmar eczema as defined by the Danish Contact Dermatitis Group
* Patients with predominantly atopic dermatitis, in which the hands are also involved. Patients with mild atopic dermatitis, in which the hands are mainly affected are eligible for inclusion.
* Psoriasis
* Active bacterial, fungal, or viral infection of the hands
* Pregnant/lactating or planning to become pregnant during the study period
* Treatment with systemic medication or UV radiation within the previous 4 weeks
* Mentally incompetent
* Immunocompromised status
* Known or suspected allergy to ingredients in the study medications
* Inclusion in a study of an investigational drug within 60 days prior to start of treatment
* Current malignancy (other than successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and⁄or localized carcinoma in situ of the cervix)
* Current active pancreatitis
* Living vaccine (including bacillus Calmette-Guérin (BCG), varicella, measles, mumps, rubella, yellow fever, oral polio and oral typhoid) in the last 2 weeks or the planned application of such a vaccine during the study period
* Evidence of alcohol abuse or drug addiction
* Chronic or recurrent infectious diseases
* Contact sensitizations with clinical relevance to the hands, in which exposure to allergens is not avoided
* Hypervitaminosis A due to the use of vitamin A supplements containing >2000 IU
* Use of drugs with potential to change the effective dosis of study drugs within the previous 2 weeks

Laboratory exclusion criteria post randomization

* Alanine aminotransferase (ALAT) and ⁄or aspartate aminotransferase (ASAT) values > 200% of the upper limit of normal
* Impaired renal function as indicated by a clinically relevant abnormal creatinine value (to be determined by investigator or treating physician)
* Anemia as indicated by a clinically relevant lowered hemoglobin value (to be determined by investigator or treating physician)

Alitretinoin specific

* Triglycerides > 200% of the upper limit of normal,
* Cholesterol or low density lipoprotein (LDL) cholesterol values > 200% of the upper limit of normal
* Uncontrolled hypothyroidism (to be determined by investigator or treating physician)

Azathioprine specific

• Patients with low or absent thiopurine methyltransferase (TPMT) activity (defined in our center as <52 nmol/gHb/hour, combined with genotyping showing homozygous of compound heterozygous mutations) and a subsequent risk for life-threatening myelotoxicity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Response to treatment/hand eczema severity (Photoguide) | 24 weeks (end of treatment)

SECONDARY OUTCOMES:
Response to treatment/hand eczema severity (Photoguide) | 12 weeks
Response to treatment/hand eczema severity (Hand Eczema Severity Index, HECSI) | Week 4, 8, 12, 24
Time to response | Week 4, 8, 12, 24
Patient reported improvement (Patient Global Assessment, PaGA) | Week 12 and 24
Safety and tolerability (adverse events) | Up to 24 weeks
Cost-utility. QALY's: registered direct/indirect costs, combined with EQ-5D outcome | Week 12 and 24
Cost-effectiveness: registered direct/indirect costs combined with the primary and secondary effectiveness outcomes (Photoguide/HECSI) | Week 12 and 24
Quality of Life: questionnaire. | Week 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: MLA Schuttelaar, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will be published anonymously and will not be possible to trace back to individual participants.